CLINICAL TRIAL: NCT04711720
Title: A Randomized Controlled, Multicenter Study for Patients Underwent Total Hip Arthroplasties Assisted by "VTS"Surgical Navigation System
Brief Title: A Randomized Controlled Trial for Patients Underwent Total Hip Arthroplasties Assisted by Surgical Navigation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Qianfoshan Hospital (Other); Chifeng Municipal Hospital (Other); Jining Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTSTH
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation (Experimental)
  Interventions: Device: "VTS" surgical navigation system
- Control (No Intervention)

INTERVENTIONS:
Device: "VTS" surgical navigation system — The"VTS" surgical navigation system can accurately match the preoperative and intraoperative image data with the patient's anatomical structure on the operating table, track the surgical instruments during the operation, and update the position of the surgical instruments on the patient's image in real time, so that the doctor can clearly understand the position of the surgical instruments relative to the patient's anatomical structure, and make the operation procedure more accurate and safer.
  Arms: Navigation

SUMMARY:
This is a randomized controlled, multicenter study. According to the inclusion criteria, volunteers were recruited from patients undergoing total hip arthroplasty. After signing the informed consent, the subjects were assigned to the experimental group and the control group through the central randomization system. The researchers will complete the total hip arthroplasty for patients in the experimental group with the assistance of surgical navigation system. The patients in the control group do not use the surgical navigation system. The proportion of acetabular abduction angle and anteversion angle in the lewinnek safe area is the primary outcome measurement. The operation time, WOMAC score, Harris score, range of motion and dislocation rate are the secondaryoutcome measurements. The incidence of complications, devices and other adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of primary hip osteoarthritis(OA), fracture of femoral neck (FFN),or secondary hip osteoarthritis due to developmental dysplasia of the hip (DDH), hip avascular necrosis (AVN), rheumatoid arthritis (RA), ankylosing spondylitis (AS), and coxa plana

Exclusion Criteria:

Severe vascular diseases of the lower extremity Neuromuscular diseases Infectious diseases Severe dysfunctions of major organs Severe neurosensory deficiencies caused by spinal diseases Unable to receive CT/MRI scans

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Acetabular location accuracy | Within 1 week after surgery
  Proportion of abduction angle and anteversion angle of acetabular cup in lewinnek safe area

SECONDARY OUTCOMES:
Operation time | Immediately after surgery
  Time from skin incision to wound closure
the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months after surgery
  The WOMAC is a self administered questionnaire to assess joint function and quality of life for patients with osteoarthritis; it consists of 24 items: pain (5 items), stiffness (2 items), and physical function (17 items). The higher the total score, the worse the patient's pain, stiffness, and functional limitations. The WOMAC is validated for various languages, including Chinese
Harris Hip Score (HHS) | 6 months after surgery
  a rating scale with a maximum of 100 points, including the domains of pain, function, deformity, and motion

IPD SHARING:
Plan to Share IPD: No